CLINICAL TRIAL: NCT00782938
Title: Serum Anticholinergic Activity (SAA) and BIS-EEG as Potential Markers for Cognitive Ability and/or the Anticholinergic Medication in ACVB Patients
Brief Title: The Role of Serum Anticholinergic Activity in ACVB Patients
Status: Completed | Type: Observational
Sponsor: Heidelberg University (Other)
Responsible Party: Plaschke, Konstanze, Department of Anesthesiology
Other Study IDs: S235-2008
Record Dates: First submitted 2008-10-30; First posted 2008-10-31 (Estimated); Last update posted 2010-01-14 (Estimated); Status verified 2008-10

CONDITIONS: Acetylcholine; Cognition; BIS-EEG

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- low SAA
- high SAA

SUMMARY:
Drugs with anticholinergic potential increase the risk of postoperative transient and persistent cognitive dysfunction especially in cardiac patients. The investigators main goal is to identify preoperative risk factors and to monitor postoperative patients' state in relation to SAA activity and bilateral BIS-EEG changes.

ELIGIBILITY:
Inclusion Criteria:

* written compliance to the study participation
* a good knowledge in German speech
* no red/ green blindness
* no previous neurological and/or psychiatric illness
* good ability to see and to hear
* Mini-Mental-State-Examination (MMSE) better than 25 points

Exclusion Criteria:

* no written compliance to the study participation
* bad knowledge in German speech
* red/ green blindness
* previous neurological and/or psychiatric illness
* no ability to see and to hear
* Mini-Mental-State-Examination (MMSE) lower than 25 points

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ACVB patients:
  Ages Eligible for Study: 55 years to 90 years Genders Eligible for Study: Both Accepts Healthy Volunteers: No
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2008-05; Primary Completion 2009-12 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Cognitive dysfunction measured by neurocognitive test battery | 3 month postsurgery

SECONDARY OUTCOMES:
SAA, BIS-EEG, descriptive patients' characteristics | 24 h postsurgery

CONTACTS AND LOCATIONS:
Overall Officials: Eike Martin, Prof., Study Chair — Department of Anesthesiology, University of Heidelberg
Locations (1):
- University of Heidelberg, Department of Anesthesiology, Heidelberg Medical School, Heidelberg, Baden-Wurttemberg, Germany

REFERENCES:
- See also: ISPOCD1 study — http://www.ncbi.nlm.nih.gov/sites/entrez